CLINICAL TRIAL: NCT01109147
Title: Comparison of the Effects of Aripiprazole and Risperidone on the Pattern of Brain Activation in Schizophrenic Patients During Emotional Tasks and With Reference to Controls
Brief Title: Comparison of the Effects of Aripiprazole and Risperidone on the Pattern of Brain Activation in Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qualissima (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009-017673-38
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia, Undifferentiated Type
Keywords: Schizophrenic Disorders; Schizophrenia; Affect; Emotional Blunting
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- aripiprazole (Active Comparator): Imagery: A fMRI session is conducted on schizophrenic patients under aripiprazole (medication taken and stabilized for at least six weeks before inclusion, no intervention on the medication is scheduled during the study).
  Genetic: pharmacogenetic sampling. One sample was collected for each subject.
  Interventions: Other: Imagery; Genetic: pharmacogenetic sampling
- risperidone (Active Comparator): Imagery: A fMRI session is conducted on schizophrenic patients under rsiperidone (medication taken and stabilized for at least six weeks before inclusion, no intervention on the medication is scheduled during the study).
  Genetic: pharmacogenetic sampling. One sample was collected for each subject.
  Interventions: Other: Imagery; Genetic: pharmacogenetic sampling
- control (Other): Imagery: A fMRI session is conducted on healthy volunteers. Genetic: pharmacogenetic sampling. One sample was collected for each subject.
  Interventions: Other: Imagery; Genetic: pharmacogenetic sampling

INTERVENTIONS:
Other: Imagery — All the subject will be submitted to an functional magnetic resonance imaging (fMRI) examination.
Genetic: pharmacogenetic sampling — A pharmacogenetic sample will be done with an additional consentment.

SUMMARY:
After an initial screening visit, including an assessment of psychiatric disorders, patients stabilized on antipsychotic medication (aripiprazole or risperidone) for at least 6 weeks and control subjects will undergo an assessment using functional magnetic resonance imaging (fMRI) of the differences of patterns of brain activation during an emotional task

DETAILED DESCRIPTION:
This study is: interventional, comparative, open label, multi center, without experimental treatment.

Main objective: To evaluate the effect of aripiprazole and risperidone on brain activation during an emotional task of matching patients with schizophrenia, and in reference to control subjects.

Secondary Objective: Comparison of emotional subjective and physiological perception in patients with schizophrenia in relation with their treatment. Comparison of brain activation in patients during the emotional induction task based on symptomatic dimensions, personality traits and performance on cognitive and attentional tests, and for insight capacity . Comparison of transcript level of candidate genes in blood mononuclear cells between the study groups and study the interactions between the observed differences in brain imaging and different levels of transcription of these genes.

ELIGIBILITY:
Inclusion Criteria:

* For patients

  1. Men and women, right handed, 18 to 45 years;
  2. Having given their written informed consent;
  3. Presenting a diagnosis of schizophrenia made by DMS IV, hospitalized or followed regularly in a hospital proper, and whose symptoms are stable for at least 6 weeks, at the discretion of the psychiatrist;
  4. Receiving antipsychotic treatment (risperidone or aripiprazole) monotherapy stable (treatment and dose) for at least than 6 weeks;
  5. Showing no contra-indication for fMRI;
  6. Patients whose physical examination is unremarkable clinically significant;
  7. Patients without serious somatic pathology;
  8. Affiliated to a social security system.
  9. For women of childbearing potential, an appropriate contraception is mandatory and an negative pregnancy test
* For controls

  1. Men and women, right handed, aged 18 to 45 years of age, sex and socio-educational level comparable to patients included;
  2. Having given their written informed consent;
  3. Do not present a diagnosis of schizophrenia according to DSM IV set;
  4. Do not present psychiatric history, and free of any psychotropic medication;
  5. Including the physical examination is unremarkable clinically significant;
  6. Having no professional musical practice;
  7. Affiliated with a social security system.

Exclusion Criteria:

* For patients

  1. Patients in menstruation without effective contraception (oral, intramuscular hormonal, intrauterine device, or surgical);
  2. Patients who are pregnant or breastfeeding;
  3. Patients not meeting criteria for schizophrenia according to DSM IV criteria or those with resistant schizophrenia (Kane criteria);
  4. Introducing a somatic disease or serious neurological, particularly Parkinson's disease, epilepsy, tardive dyskinesia and disabling cardiovascular disease, liver or kidney disease;
  5. Presenting a contra-indication to MRI;
  6. Having a history of alcoholism or drug addiction during the past year;
  7. Participating in another clinical trial or are in a period of exclusion from a previous protocol;
  8. Patients likely to have behavioral self aggression from the trial investigators

     During the study:

  <!-- -->

  1. The investigator considers, for safety reasons, it is in the interest of the patient to be excluded from the study (Hospital readmission due to psychotic symptoms, clinical or psychiatric reasons)
  2. Consentment withdrawal
  3. The patient does not longer correspond to the inclusion criteria or protocol requirements
* For controls

  1. Women of childbearing potential without effective contraception (oral, intramuscular hormonal, intrauterine device, or surgical);
  2. Pregnant or breastfeeding;
  3. Presenting a somatic, psychiatric or neurological disorder;
  4. Presenting a history of alcohol or substance abuse during the past year;
  5. Participating in another clinical trial or are in a period of exclusion from a previous protocol;
  6. Presenting a contra-indication to MRI.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Blin, professor, Study Director — study coordinator
Locations (2):
- France (2):
  - Sainte-Marguerite Hospital - Psychiatric service -Service du Pr Azorin - 270 boulevard de Sainte Marguerite, Marseille
  - Hôpital de la Conception - Service du Pr Dassa -147, boulevard Baille, Marseille

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Schizophrenic patient stabilized under aripiprazole for six weeks before inclusion
- Risperidone: Schizophrenic patient stabilized under risperidone for six weeks before inclusion
- Control: healthy volunteers
Period: Overall Study
Arm/Group | Aripiprazole | Risperidone | Control
Started | 17 | 14 | 36
Completed | 15 (2 have been excluded of the results) | 11 (3 have been excluded of the results) | 26 (10 have been excluded of the results)
Not Completed | 2 | 3 | 10

BASELINE CHARACTERISTICS:
Population: The number of participants was calculated as an estimation, due to no previous known results in this field of research.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Risperidone | Control | Total
Number analyzed (Participants) | 17 | 14 | 36 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 36 | 67
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (9.6) | 31.6 (9.2) | 32.9 (7.8) | 33.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12 | 24
  Male | 9 | 10 | 24 | 43
Region of Enrollment [Number; unit: participants]
  France | 17 | 14 | 36 | 67

OUTCOME MEASURES:

1. Secondary Outcome: Assessment of Emotional Reactivity
Time Frame: 3 days after the decision of inclusion
Reporting Status: Not Posted

2. Secondary Outcome: Assessment of Cognitive and Attentional Abilities
Time Frame: 3 days after the decision of inclusion
Reporting Status: Not Posted

3. Secondary Outcome: Assessment of Personality Traits
Time Frame: 3 days after the decision of inclusion
Reporting Status: Not Posted

4. Secondary Outcome: Investigate the Level of Expression of Candidate Genes
Time Frame: one blood sample
Reporting Status: Not Posted

5. Primary Outcome: Identification of Brain Circuits Involved in a Task of Emotional Congruence (With fMRI)
Description: During the fMRI session, the activation of each brain circuits is measured by a "Bold signal" (an arbitrary measure of contrast: numbers of voxels highlighted/activated in the region of interest).
  The emotional task is composed by congruent and incongruent images. Three effects were caused by the task: congruence, attention and valence effects. Each of them affect, involve and activate the regions of interests differentially within the differents arms.
  The region of interests who were mainly observed are: Anterior Cingulate Cortex (ACC), Prefrontal dorso-lateral Cortex (PFdlC) and the Amygdala (A).
Time Frame: 3 days after the decision of inclusion
Measure: Mean (Standard Error); unit: arbitrary units of activation
Arm/Group | Aripiprazole | Risperidone | Control
Number analyzed (Participants) | 15 | 11 | 26
arbitrary units of activation
  Activation of Anterior Cingulate Cortex (ACC) | -0.25 (2.8) | -0.21 (3.1) | 3.8 (3.2)
  Activation of Prefrontal dorso-lateral Cortex (PF) | 0.2 (3.0) | -0.3 (4.0) | 5.3 (5.0)

ADVERSE EVENTS:
Time Frame: Assessment of adverse event at each visit (2 times on approximately one week).
Description: Assessment of adverse event has been run by the investiagtor at each visit (2 times) during the entire participation of the subject (approximately one week).
Arm/Group | Aripiprazole | Risperidone | Control
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/36
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=17) | Risperidone (N=14) | Control (N=36)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — after a blood puncture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All results and publications are reviewed by the sponsor and the principle Investigator. None could be released without accordance from both parts.